CLINICAL TRIAL: NCT05463601
Title: Efficacy and Safety of Mecapegfilgrastim for Prophylaxis of Dalpiciclib -Induced Neutropenia in Patients With Advanced HR+/HER2- Breast Cancer: a Open-label, Multicenter, Investigator-initiated, Randomized Controlled Phase II Trial
Brief Title: Mecapegfilgrastim for the Prevention of Dalpiciclib -Induced Neutropenia in Advanced Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jieqiong Liu, M.D., Ph.D., Associate Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SYSKY-2022-105-01
Record Dates: First submitted 2022-06-01; First posted 2022-07-19 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pegylated granulocyte colony-stimulating factor; dalpiciclib; exemestane; Fulvestrant; Letrozole; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mecapegfilgrastim +dalpiciclib + endocrine therapy (Experimental): Mecapegfilgrastim / dalpiciclib / Endocrine therapy (exemestane, fulvestrant, letrozole, tamoxifen)
  Interventions: Drug: Mecapegfilgrastim; Drug: dalpiciclib; Drug: exemestane, fulvestrant, letrozole, tamoxifen
- dalpiciclib + endocrine therapy (Active Comparator): dalpiciclib / Endocrine therapy (exemestane, fulvestrant, letrozole, tamoxifen)
  Interventions: Drug: dalpiciclib; Drug: exemestane, fulvestrant, letrozole, tamoxifen

INTERVENTIONS:
Drug: Mecapegfilgrastim — Mecapegfilgrastim
  Arms: Mecapegfilgrastim +dalpiciclib + endocrine therapy
Drug: dalpiciclib — dalpiciclib
Drug: exemestane, fulvestrant, letrozole, tamoxifen — endocrine therapy

SUMMARY:
Neutropenia is a common complication from dalpiciclib. Mecapegfilgramtim (code name HHPG-19K), a long-acting recombinant human granulocyte colony-stimulating factor (rhG-CSF), has been developed. The study aim to evaluate the safety and efficiency of mecapegfilgrastim for prophylaxis of dalpiciclib -induced neutropenia in patients with advanced HR+/HER2- breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18.
2. Pathologically confirmed advanced HR+/HER2- breast cancer: there is evidence of focal recurrence or metastasis, which is not suitable for surgical resection or radiotherapy for the purpose of cure.
3. No more than one line of chemotherapy is allowed for patients with recurrent and metastatic diseases.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
5. For patients with brain metastases, there is need for local treatment, and the brain lesions are stable for ≥ 3 months, and no need for dexamethasone or mannitol.
6. Adequate organ function: (I) adequate hematologic function: hemoglobin ≥90 g/L, absolute neutrophil count (ANC) ≥1.5×109/L, platelet count (PLT) ≥100×109/L; (II) adequate renal and hepatic function.
7. Negative pregnancy test.

Exclusion Criteria:

1. Previous pathological diagnosis of HER2 positive breast cancer.
2. Previous treatment with cdk4/6 inhibitors.
3. Major surgery, chemotherapy, radiotherapy, any research drug or other anti-cancer treatment within 2 weeks before entering the trial.
4. Any other malignant tumor diagnosed within 3 years before entering the study, except non-melanoma skin cancer, basal cell or squamous cell skin cancer or cervical carcinoma in situ after radical treatment.
5. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV DNA ≥ 1000 IU/ml), hepatitis C (HCV antibody positive and HCV-RNA higher than the detection limit of the analytical method) or combined hepatitis B and hepatitis C co-infection.
6. Within 6 months before entering the study, the following conditions occurred: myocardial infarction, severe / unstable angina pectoris, NYHA grade 2 or above cardiac insufficiency, persistent arrhythmia ≥ grade 2 (according to nci-ctcae version 5.0), atrial fibrillation at any level, coronary / peripheral artery bypass grafting, symptomatic congestive heart failure, cerebrovascular accident (including transient ischemic attack or symptomatic pulmonary embolism).
7. Inability to swallow, intestinal obstruction or other factors affecting drug administration and absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade ≥3 neutropenia at the end of cycle 1 (each cycle is 28 days) | at the end of cycle 1 (each cycle is 28 days)
  The incidence of grade ≥3 neutropenia in cycle 1: defined as ANC <1.0×109/L at the end of Cycle 1 (each cycle is 28 days).

SECONDARY OUTCOMES:
The incidence of grade ≥3 neutropenia at the end of all cycles (each cycle is 28 days) | through study completion, an average of 2 years
  The incidence of grade ≥3 neutropenia of all cycles: defined as ANC <1.0×109/L at the end of All Cycles (each cycle is 28 days).
Breast-Q scores | through study completion, an average of 2 years
  Breast-Q scores for patient's quality of life
Progression-free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Progression-free Survival
Overall Survival | From date of randomization until the date of death from any cause, assessed up to 60 months
  Overall Survival
Relative dose intensity of dalpiciclib | through study completion, an average of 2 years
  Relative dose intensity of dalpiciclib
Objective response rate (ORR） | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Objective response rate

CONTACTS AND LOCATIONS:
Locations (1):
- 中山大学中山纪念医院, Guangzhou, Guangdong, China